CLINICAL TRIAL: NCT02234570
Title: A Randomized, Double-Blind Placebo-Controlled Phase I Trial Evaluating the Safety and Pharmacokinetics of Oxfendazole
Brief Title: Phase I Trial Evaluating the Safety and Pharmacokinetics of Oxfendazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-0053
Record Dates: First submitted 2014-08-28; First posted 2014-09-09 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2019-12-05

CONDITIONS: Neurocysticercosis
Keywords: neurocysticercosis; pork tapeworm; Taenia solium
MeSH Terms: conditions — Neurocysticercosis; Taeniasis | interventions — oxfendazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1 (Experimental): N=8 subjects receive single oral dose 0.5mg/kg of oxfendazole; N= 2 subjects receive single oral dose placebo
  Interventions: Drug: Oxfendazole; Other: Placebo
- Group 2 (Experimental): N=8 subjects receive single oral dose 1mg/kg of oxfendazole; N=2 subjects receive single oral dose placebo
  Interventions: Drug: Oxfendazole; Other: Placebo
- Group 3 (Experimental): N=8 subjects receive single oral dose 3mg/kg of oxfendazole; N= 2 subjects receive single oral dose placebo
  Interventions: Drug: Oxfendazole; Other: Placebo
- Group 4 (Experimental): N=8 subjects receive single oral dose 7.5mg/kg of oxfendazole; N=2 subjects receive single oral dose placebo
  Interventions: Drug: Oxfendazole; Other: Placebo
- Group 5 (Experimental): N=8 subjects receive single oral dose 15mg/kg of oxfendazole; N= 2 subjects receive single oral dose placebo
  Interventions: Drug: Oxfendazole; Other: Placebo
- Group 6 (Experimental): N=8 subjects receive single oral dose 30mg/kg of oxfendazole; N=2 subjects receive single oral dose placebo
  Interventions: Drug: Oxfendazole; Other: Placebo
- Group 7 (Experimental): N=8 subjects receive single oral dose 60mg/kg of oxfendazole; N=2 subjects receive single oral dose placebo
  Interventions: Drug: Oxfendazole; Other: Placebo

INTERVENTIONS:
Drug: Oxfendazole — A benzimidazole carbamate antiparasitic drug. Oral Dose levels of 0.5,1, 3, 7.5, 15, 30, and 60 mg/kg will be evaluated sequentially, the dose increasing with each new cohort Group 1 to Group 7.
Other: Placebo — Normal Saline administered with an oral dosing syringe. Group 1- Group 6

SUMMARY:
The objectives of the Phase I study are to evaluate the safety and tolerance of increasing single oral doses of oxfendazole in healthy volunteers.The secondary objectives assess the pharmacokinetic profile of oxfendazole and assess the metabolism of oxfendazole. The description of agent used is single oral dose of an aqueous suspension of oxfendazole, a benzimidazole carbamate antiparasitic drug. Each new cohort will be dosed only after the two week safety data for the preceding group have been reviewed. If a clinically significant AE is observed, and if this event is drug-related the safety monitoring committee will be convened to determine whether the study should continue.

DETAILED DESCRIPTION:
This Phase I study is a randomized, double-blind, placebo-controlled evaluation of the safety and pharmacokinetics of escalating single oral doses of oxfendazole (0.5 to 60 mg/kg) in healthy volunteers. Up to 70 healthy males and females (non-chldbearing potential), ages 18-45 volunteers recruited from one site will participate in this study. The study duration is approximately 18 months with subject participation of 2 weeks. The primary objective assess the safety and tolerability of oxfendazole in healthy adults. The secondary objectives assess the pharmacokinetic profile of oxfendazole and assess the metabolism of oxfendazole. Two sentinel subjects will receive the study product (1 drug/1 placebo) in each group and be monitored 48 hours for adverse events prior to completing enrollment of the remaining 8 subjects in the group.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of non-childbearing potential between the ages of 18 and 45 years, inclusive.* *Surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who have been postmenopausal for >/=1 year confirmed by LH and FSH levels. 2. In good health, as judged by the investigator and determined by vital signs* Temperature < 38 degrees Celsius, heart rate </=100 bpm and > 50 bpm, systolic blood pressure </= 140 mmHg and > 89 mmHg, diastolic blood pressure </=90 mmHg and >/= 60 mm Hg, medical history and a targeted physical examination. BMI >/=18 and </= 35. Athletically trained subjects with a pulse >/= 45 may be enrolled at the discretion of the principal investigator or designated licensed clinical investigator. 3. Acceptable screening laboratories* *Hemoglobin, white blood cell (WBC) count, neutrophil, eosinophil and platelet counts within normal ranges. AST < 44 and ALT < 44 and total bilirubin, creatinine must be equal to or below the upper limit of normal (for eosinophil count, AST, ALT, creatinine, and total bilirubin values below the normal range are acceptable). Random blood glucose must be <140. Urine dipstick testing must be negative for glucose and negative or trace for protein. The following serology tests must be negative: HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody. HIV and hepatitis C viral load PCR testing may be performed for individuals suspected of having indeterminate antibody testing. 4. Male participants must be willing to ensure use of condoms and spermicides for 4 months after study drug administration. 5. Provide written informed consent before initiation of any study procedures. 6. Willing to be available for all study-required procedures, and visits for the duration of the study. 7. Able to provide a home phone number, and the name, address, and/or email of a person willing to assist with making contact during the follow-up phase of the study.

Exclusion Criteria:

1. History of residing for 6 or more months in regions with endemic cysticercosis as determined by the principal investigator or a designated study physician. 2. Breastfeeding females. 3. Body temperature >/=100.4 degrees Fahrenheit (>/=38.0 degrees Celsius) or acute illness within 3 days before administration of study drug (subject may be rescheduled). 4. Chronic or acute medical disorder* *Disorders of the cardiac, pulmonary, liver, kidney, neurologic, gastrointestinal or other system, such that in the opinion of the investigator participation in the study creates additional risk to the subject, or to the validity of the study. 5. Use of chronic systemic medications* *Intermittent use of over the counter medications such as acetaminophen, ibuprofen, cold and sinus medications are permitted for enrollment (please see section 5.6 for instructions on medication use during the study).Topical medications, nasal steroids are permitted throughout the study. Use of the prescription medications used less than once per week on average are permitted for enrollment (see section 5.6 for instructions on medication use during the study). If the subject has taken a short term prescription medication within the past 30 days (e.g. an antibiotic), they should be postponed from enrollment until 30 days have elapsed since the last dose 6. Has history of sensitivity to related benzimidazole compounds (e.g., albendazole, mebendazole). 7. A diagnosis of schizophrenia, bipolar disease, or history of hospitalization for a psychiatric condition or previous suicide attempt. 8. A history of treatment for any other psychiatric disorder in the past 3 years.* *Past treatment for ADHD does not exclude participants from enrollment as long as the medications have been discontinued for a minimum of 3 months and symptoms are well controlled. 9. Received an experimental agent* within 1 month before administration of study drug or expect to receive an experimental agent during the 15-day study period. *Vaccine, drug, biologic, device, blood product, or medication. 10. Any condition that would, in the opinion of the investigator, place them at an unacceptable risk of injury, render them unable to meet the requirements of the protocol, or that may interfere with successful completion of the study. 11. A history of alcohol consumption* or any illicit drug use†, or history of substance abuse#. Individuals must agree to abstain from drug or alcohol use for 48 hours prior to enrollment through day 15. *Greater than 7 alcoholic drinks per week. †Other than occasional marijuana use (less than once per week for the past 60 days is acceptable). #Alcohol or illicit drugs within the past 3 years. 12. History of chronic tobacco use in the past 60 days.* *A history of occasional tobacco use (less than 1 pack per week on average) is acceptable. Individuals will be counseled to abstain from use of tobacco and marijuana from screening through day 15.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2015-11-24 (Actual); Study Completion 2015-11-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa, United States

REFERENCES:
- [Derived] An G, Murry DJ, Gajurel K, Bach T, Deye G, Stebounova LV, Codd EE, Horton J, Gonzalez AE, Garcia HH, Ince D, Hodgson-Zingman D, Nomicos EYH, Conrad T, Kennedy J, Jones W, Gilman RH, Winokur P. Pharmacokinetics, Safety, and Tolerability of Oxfendazole in Healthy Volunteers: a Randomized, Placebo-Controlled First-in-Human Single-Dose Escalation Study. Antimicrob Agents Chemother. 2019 Mar 27;63(4):e02255-18. doi: 10.1128/AAC.02255-18. Print 2019 Apr. PMID 30745383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult males and non-pregnant females recruited from existing volunteer populations and from the communities at large around the clinical site. Participants were enrolled between 17NOV2014 and 09NOV2015.
Groups:
- 0.5 mg/kg Oxfendazole: Participants received a single oral dose 0.5 mg/kg of oxfendazole.
- 1 mg/kg Oxfendazole: Participants received a single oral dose 1 mg/kg of oxfendazole
- 3 mg/kg Oxfendazole: Participants received a single oral dose 3 mg/kg of oxfendazole
- 7.5 mg/kg Oxfendazole: Participants received a single oral dose 7.5 mg/kg of oxfendazole
- 15 mg/kg Oxfendazole: Participants received a single oral dose 15 mg/kg of oxfendazole
- 30 mg/kg Oxfendazole: Participants received a single oral dose 30 mg/kg of oxfendazole
- 60 mg/kg Oxfendazole: Participants received a single oral dose 60 mg/kg of oxfendazole
- Placebo: Participants received a single placebo formulation consisting of 4.5% polyethylene glycol, 0.18% methyl paraben, and 95.32% sterile water for injection
Period: Overall Study
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole | Placebo
Started | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 14
Completed | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants are included in the analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 14 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 14 | 70
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (6.7) | 26.6 (6.8) | 23.8 (6.1) | 26.3 (7.1) | 26.8 (9.3) | 22.6 (6.7) | 24.6 (8.0) | 26.9 (7.2) | 25.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3
  Male | 8 | 7 | 8 | 7 | 8 | 8 | 8 | 13 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 0 | 2 | 1 | 2 | 0 | 8
  Not Hispanic or Latino | 8 | 7 | 5 | 8 | 6 | 7 | 6 | 14 | 61
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 4
  White | 7 | 8 | 7 | 6 | 5 | 6 | 6 | 12 | 57
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 14 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Adverse Events Related to Oxfendazole Within 14 Days of Receipt of a Single Oral Dose.
Description: All adverse events, defined as any untoward medical occurrence regardless of its causal relationship to the study treatment, were collected for 14 days after dosing. The PI then determined relatedness to the study drug. Related was defined as "there is a reasonable possibility that the study product caused the adverse event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the adverse event."
Time Frame: Within 14 Days of first dose
Population: All participants are included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 14
Participants | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1

2. Secondary Outcome: Area Under the Concentration Time-curve From Time Zero to Infinity (AUC(0-infinity)) for Oxfendazole
Description: AUC(0-infinity) was defined as the total area under the concentration-time curve from dosing (time 0) taken to the limit as the end time becomes arbitrarily large. AUC(0-infinity) and was calculated by adding AUC(0-last) to an extrapolated value equal to the last measured concentration greater than the lower limit of quantification of the bioanalytical assay divided by the terminal phase elimination rate constant (Ke) computed from concentrations that were measured using a validated HPLCMS/MS method
Time Frame: 0, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 336 hours post-dose
Population: All participants receiving oxfendazole are included in the analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
ng•hr/mL | 11682.4 (44.8) | 13117.7 (54.4) | 30803.1 (20.1) | 73928.9 (40.6) | 99542.6 (23.9) | 78344.0 (34.4) | 108618.2 (38.4)

3. Secondary Outcome: Maximum Observed Concentration (Cmax) of Oxfendazole in Plasma
Description: Cmax is defined as the maximum observed drug concentration observed in plasma over all PK sample concentrations computed from concentrations that were measured using a validated HPLC-MS/MS method.
Time Frame: 0, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 336 hours post-dose
Population: All participants receiving oxfendazole are included in the analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
ng/mL | 943.9 (28.4) | 1155.9 (26.8) | 2436.9 (24.0) | 4781.3 (25.6) | 6254.8 (21.7) | 5301.3 (30.5) | 6768.4 (31.3)

4. Secondary Outcome: Plasma Concentrations of Oxfendazole Fenbendazole
Description: Concentrations of oxfendazole fenbendazole in plasma were measured using a validated HPLCMS/MS method. Concentrations <LLOQ (2 ng/mL) set to LLOQ/2 if after 1st =LLOQ concentration or 0 otherwise for calculating summary statistics.
Time Frame: Day 1-Day15
Population: All participants receiving oxfendazole are included in the analysis population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
ng/mL
  1 Hour | 0 (0) | 0 (0) | 0.3 (0.8) | 0.3 (0.7) | 1.0 (1.4) | 1.4 (1.2) | 5.9 (2.4)
  2 Hours | 0 (0) | 0 (0) | 0.4 (0.8) | 1.1 (1.5) | 2.6 (2.5) | 2.2 (1.5) | 6.3 (2.5)
  4 Hours | 0.6 (1.8) | 0.8 (1.1) | 3.5 (2.5) | 3.0 (3.2) | 8.1 (8.0) | 4.4 (4.3) | 8.0 (3.6)
  6 Hours | 0.5 (1.3) | 2.0 (1.4) | 4.8 (2.9) | 6.6 (4.8) | 9.9 (8.3) | 5.8 (6.7) | 12.4 (4.9)
  8 Hours | 0.3 (0.9) | 1.9 (1.2) | 5.2 (2.9) | 6.7 (4.6) | 10.8 (8.3) | 5.0 (5.1) | 15.5 (8.6)
  10 Hours | 0.3 (0.8) | 2.3 (1.2) | 6.8 (2.6) | 10.0 (5.7) | 11.2 (6.6) | 5.5 (4.5) | 18.4 (11.1)
  12 Hours | 0.3 (0.9) | 2.3 (1.4) | 6.7 (2.4) | 10.1 (5.5) | 11.7 (7.9) | 6.4 (4.5) | 20.9 (19.0)
  24 Hours | 0.7 (1.0) | 2.3 (1.6) | 7.1 (2.5) | 4.9 (4.0) | 10.0 (3.7) | 5.4 (3.2) | 16.7 (12.9)
  Day 3 | 0.4 (0.5) | 0.9 (0.4) | 3.2 (2.8) | 2.2 (1.7) | 3.7 (3.4) | 2.5 (3.1) | 5.5 (4.2)
  Day 4 | 0.4 (0.5) | 0.9 (0.4) | 1.1 (0.4) | 1.4 (1.0) | 1.2 (0.6) | 1.3 (1.4) | 2.5 (3.0)
  Day 6 | 0.4 (0.5) | 0.9 (0.4) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 0.9 (0.4) | 1.7 (1.9)
  Day 8 | 0.4 (0.5) | 0.9 (0.4) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 0.9 (0.4) | 1.0 (0.0)
  Day 15 | 0.4 (0.5) | 0.9 (0.4) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 0.9 (0.4) | 1.0 (0.0)

5. Secondary Outcome: Plasma Concentrations of Oxfendazole Sulfone
Description: Concentrations of oxfendazole sulfone in plasma were measured using a validated HPLCMS/MS method. Concentrations <LLOQ (2 ng/mL) set to LLOQ/2 if after 1st =LLOQ concentration or 0 otherwise for calculating summary statistics.
Time Frame: Day 1-Day15
Population: All participants receiving oxfendazole are included in the analysis population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
ng/mL
  1 Hour | 28.5 (4.6) | 31.1 (11.1) | 73.0 (24.1) | 100.5 (25.4) | 111.6 (51.9) | 161.5 (41.3) | 209.1 (84.5)
  2 Hours | 48.7 (9.3) | 56.0 (11.3) | 106.3 (31.5) | 182.3 (51.6) | 219.2 (73.0) | 262.6 (72.5) | 319.0 (119.9)
  4 Hours | 52.3 (8.6) | 67.6 (16.0) | 108.1 (25.7) | 223.8 (62.5) | 258.6 (73.0) | 285.7 (74.5) | 345.4 (133.0)
  6 Hours | 57.3 (15.1) | 75.1 (26.6) | 113.8 (26.2) | 264.1 (63.0) | 308.3 (98.8) | 330.3 (90.1) | 404.6 (154.7)
  8 Hours | 59.7 (13.7) | 78.2 (27.0) | 135.5 (33.9) | 296.2 (71.5) | 336.8 (72.2) | 356.3 (120.1) | 454.8 (174.0)
  10 Hours | 62.8 (22.3) | 70.7 (28.5) | 119.4 (18.7) | 308.7 (120.1) | 340.8 (68.1) | 352.4 (106.0) | 470.7 (182.5)
  12 Hours | 56.8 (17.5) | 65.4 (30.9) | 111.4 (12.4) | 296.0 (90.3) | 359.3 (102.1) | 343.7 (111.7) | 487.7 (210.3)
  24 Hours | 30.9 (23.4) | 38.9 (31.7) | 68.5 (21.0) | 176.7 (125.5) | 261.8 (83.4) | 185.2 (90.5) | 362.2 (222.7)
  Day 3 | 11.4 (11.8) | 11.1 (10.3) | 20.8 (12.2) | 64.8 (94.9) | 75.1 (47.6) | 57.5 (54.4) | 119.5 (86.8)
  Day 4 | 3.6 (3.1) | 2.8 (3.5) | 5.7 (3.8) | 17.3 (27.2) | 16.7 (15.1) | 17.2 (23.6) | 33.8 (28.6)
  Day 6 | 1.2 (0.4) | 1.3 (1.0) | 1.3 (0.8) | 6.4 (10.2) | 1.2 (0.6) | 4.0 (7.7) | 6.6 (9.4)
  Day 8 | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.1 (0.4)
  Day 15 | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0)

6. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Oxfendazole
Description: The apparent terminal elimination half-life (t1/2) was defined as the time required for the drug concentration to decrease by a factor of one-half in the terminal phase computed from concentrations that were measured using a validated HPLCMS/MS method.
Time Frame: 0, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 336 hours post-dose
Population: All participants receiving oxfendazole are included in the analysis population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
hours | 9.1 (27.5) | 8.5 (25.3) | 10.3 (35.7) | 9.6 (34.2) | 10.0 (21.8) | 9.8 (33.7) | 11.0 (44.5)

7. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of Oxfendazole
Description: Tmax was defined as the time at which the maximum concentration (Cmax) occurs in plasma computed from concentrations that were measured using a validated HPLCMS/MS method.
Time Frame: 0, 1, 2, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 336 hours post-dose
Population: All participants receiving oxfendazole are included in the analysis population.
Measure: Median (Full Range); unit: hours
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
hours | 2.0 [2.0 to 2.1] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0] | 2.0 [2.0 to 9.5] | 2.0 [1.9 to 6.0] | 2.0 [1.4 to 7.9]

8. Secondary Outcome: Urine Concentrations of Oxfendazole Fenbendazole
Description: Concentrations of oxfendazole fenbendazole in urine were measured using a validated HPLCMS/MS method. Concentrations <LLOQ (2 ng/mL) set to LLOQ/2 if after 1st =LLOQ concentration or 0 otherwise for calculating summary statistics.
Time Frame: Day 1-Day 15
Population: All participants receiving oxfendazole are included in the analysis population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
ng/mL
  0-4 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  4-8 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  8-12 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  12-24 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  24-32 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0.03 (0.07)
  48-60 hours | 0 (0) | 0 (0) | 0 (0) | 0.28 (0.78) | 0 (0) | 0 (0) | 0 (0)

9. Secondary Outcome: Urine Concentrations of Oxfendazole Sulfone
Description: Concentrations of oxfendazole sulfone in urine were measured using a validated HPLCMS/MS method. Concentrations <LLOQ (2 ng/mL) set to LLOQ/2 if after 1st =LLOQ concentration or 0 otherwise for calculating summary statistics.
Time Frame: Day 1-Day 15
Population: All participants receiving oxfendazole are included in the analysis population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8
ng/mL
  0-4 hours | 9.1 (16.8) | 4.1 (11.6) | 19.9 (25.7) | 45.6 (37.0) | 46.4 (20.9) | 68.0 (21.2) | 64.5 (44.5)
  4-8 hours | 18.9 (13.8) | 24.9 (18.3) | 38.2 (20.3) | 86.0 (68.9) | 88.1 (27.6) | 105.8 (36.4) | 124.1 (72.8)
  8-12 hours | 34.1 (50.3) | 26.5 (22.9) | 30.3 (14.7) | 76.0 (60.1) | 92.3 (33.3) | 99.7 (40.8) | 92.9 (39.7)
  12-24 hours | 18.9 (29.1) | 26.3 (33.7) | 15.8 (18.5) | 100.4 (87.2) | 91.8 (46.7) | 69.9 (49.0) | 139.0 (137.7)
  24-32 hours | 0 (0) | 0.9 (2.6) | 1.2 (3.4) | 3.2 (4.9) | 7.5 (9.1) | 18.2 (32.4) | 26.1 (32.4)
  48-60 hours | 0 (0) | 0 (0) | 0 (0) | 0.8 (1.6) | 0 (0) | 7.3 (9.7) | 5.3 (7.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of receipt of study drug on Day 1 through approximately 14 days after receipt of study product.
Arm/Group | 0.5 mg/kg Oxfendazole | 1 mg/kg Oxfendazole | 3 mg/kg Oxfendazole | 7.5 mg/kg Oxfendazole | 15 mg/kg Oxfendazole | 30 mg/kg Oxfendazole | 60 mg/kg Oxfendazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/14
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8 | 2/8 | 0/8 | 1/8 | 1/8 | 2/8 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 mg/kg Oxfendazole (N=8) | 1 mg/kg Oxfendazole (N=8) | 3 mg/kg Oxfendazole (N=8) | 7.5 mg/kg Oxfendazole (N=8) | 15 mg/kg Oxfendazole (N=8) | 30 mg/kg Oxfendazole (N=8) | 60 mg/kg Oxfendazole (N=8) | Placebo (N=14)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram PR Prolongation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT02234570/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT02234570/SAP_001.pdf